CLINICAL TRIAL: NCT06673511
Title: A Single-Arm, Open, Multicenter, Exploratory Clinical Study on the Application of Sentinel Lymph Node Mapping Mechnique in the Surgery of Early Epithelial Ovarian Cancer
Brief Title: The Application of Sentinel Lymph Node Mapping Technique in the Surgery of Early Epithelial Ovarian Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shen zhen 2024-06
Record Dates: First submitted 2024-10-14; First posted 2024-11-05 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Epithelial Ovarian Cancer; Sentinel Lymph Node Detection
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lymph node developing group (Experimental): After injecting IGG intraoperatively, the developing lymph nodes and systemic lymph nodes are resected.
  Interventions: Procedure: Lymph node visualization
- lymph node non-developing group (Experimental): After injecting IGG intraoperatively, the developing lymph nodes and systemic lymph nodes are resected
  Interventions: Procedure: No visualization of lymph nodes

INTERVENTIONS:
Procedure: Lymph node visualization — Resect the developing lymph nodes and the systematic lymph nodes. Conduct postoperative follow-up and pay attention to the relevant indicators of the patient after surgery.
  Arms: Lymph node developing group
Procedure: No visualization of lymph nodes — Resect the systematic lymph nodes. Conduct postoperative follow-up and pay attention to the relevant indicators of the patient after surgery.
  Arms: lymph node non-developing group

SUMMARY:
This study is a single-arm, open, multicenter, exploratory clinical study to evaluate the feasibility, sensitivity, and specificity of sentinel lymph node (SLN) mapping technology in the population with early epithelial ovarian cancer in China. Patients with stage I-II epithelial ovarian cancer evaluated by preoperative imaging (enhanced CT and/or magnetic resonance scanning) are selected as the study population. The feasibility and value of SLN mapping technology in early epithelial ovarian cancer are explored through the location and number of sentinel lymph nodes, lymph node metastasis rate, 3-year disease-free survival rate, and the incidence of postoperative lower limb edema. The study plans to recruit 246 subjects. All subjects will receive study treatment after signing the informed consent form and passing the screening.

DETAILED DESCRIPTION:
This clinical study is an evaluation of surgical method improvement. The standard surgical procedure includes: selecting patients who meet the inclusion criteria, completing preoperative examinations, having thorough preoperative communication, determining laparoscopic surgery and open surgery according to the patient's condition and examinations, mainly using open surgery and strictly screening laparoscopic surgery; carefully exploring the pelvic and abdominal peritoneum and the surface of abdominal organs during the operation, evaluating whether there is lymph node enlargement in the retroperitoneum, taking ascites or peritoneal lavage fluid, after removing the patient's adnexa, sending it for rapid pathology. After the pathology is confirmed to be epithelial cancer, select a fine needle to inject 2 ml of ICG (1.25 mg/ml) respectively into the residual end of the suspensory ligament and proper ligament of the affected side. If there are lesions on both adnexa, inject on both sides; open the retroperitoneum and open the peritoneum upward to reach the level of the left renal vein; observe the lymphatic drainage area, separate the lymph and adipose tissue along the blood vessels, and look for the visualized lymph nodes; send the resected visualized lymph nodes for intraoperative rapid pathology; after resecting the visualized sentinel lymph nodes, perform systematic lymph node resection (including the para-aortic lymph nodes below the left renal vein and bilateral pelvic lymph nodes); resect the greater omentum, perform biopsy and/or resect any suspicious lesions, and perform random biopsy of normal peritoneum; resect the total uterus and suture the vaginal stump; conduct postoperative follow-up and collect statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Epithelial ovarian cancer evaluated as stage I-II by preoperative imaging (enhanced CT and/or magnetic resonance scanning), without retroperitoneal lymph node enlargement or with lymph node enlargement having a short diameter less than 1 cm.
2. Age between 18 and 75 years old (≥18 and ≤75).
3. ECOG score: 0 - 1.
4. Patients with appropriate bone marrow hematopoiesis function, renal function and liver function: white blood cell count > 3.0 x 109 cells/L; platelet count > 100 x 109/L; creatinine < 180 μmol/L; bilirubin < 1.5 times normal; aspartate aminotransferase/alanine aminotransferase < 3 times normal.
5. No fertility requirement.
6. Have signed the informed consent form.

Exclusion Criteria:

1. Advanced epithelial ovarian cancer or retroperitoneal lymph node metastasis evaluated by preoperative imaging (enhanced CT and/or magnetic resonance scanning).
2. Previous history of resection or sampling of para-aortic and/or iliac vascular lymph nodes.
3. Previous history of abdominal aorta and/or iliac vascular surgery.
4. Previous allergy to indocyanine green or iodine.
5. Previous history of abdominal radiotherapy.
6. Pregnant and lactating patients.
7. Those who refuse to sign the informed consent form.
8. Those who are considered by the investigator as inappropriate to participate in this trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | three years
  Progression-Free Survival (PFS) is defined as the time interval between the patient's diagnosis of gynecological malignancy and the first occurrence of progression of the disease or death from any cause.

SECONDARY OUTCOMES:
OS | three years
  Overall Survival (OS) was defined as the time interval between the patient's diagnosis of gynecologic malignancy and death from any cause or the end of the last follow-up date.